CLINICAL TRIAL: NCT01164969
Title: Multi Locus Sequence Typing (MLST) Used as Tool to Confirm Ability of Susceptible Helicobacter Pylori Strains to Gain Resistance to Clarithromycin During Eradication Therapy Independently of Mixed Strain Helicobacter Pylori Infection
Brief Title: Mixed Strain H. Pylori Infection in Patients Who Have Problems With Eradication of H. Pylori
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Institute of microbiology and immunology, Slovenia (Unknown)
Responsible Party: Institute of microbiology and immunology, Slovenia
Other Study IDs: IMI2010-2
Record Dates: First submitted 2010-07-13; First posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: H. Pylori Eradication Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Isolated PBMC cell from patients, isolated H. pylori
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- H. pylori eradication failure: People who are not able to eradicate H. pylori although the appropriate antibiotic therapy taken.
  Interventions: Drug: Antibiotics to which H. pylori can not develope resistance

INTERVENTIONS:
Drug: Antibiotics to which H. pylori can not develope resistance — Amoxicillin, metronidazole and tetracyclin as primary drugs to treat H. pylori infection in duration of 10 days.

SUMMARY:
The purpose of this study is to determine whether mixed H. pylori strain infection is the reason for eradication failure during treatment of H. pylori infection. The investigators present the results got from extensive sampling of biopsy samples taken from individuals diagnosed with H. pylori connected disease. The investigators were looking for individuals that were not able to eradicate H. pylori although they had susceptibility testing tailored antibiotic therapy. On their control visit after 2 months they presented again with H. pylori although at their first visit they had H. pylori isolated from biopsy sample sensitive to all antibiotics prescribed. Multi Locus Sequence Typing (MLST) was used to prove the sequence type of H. pylori and E test was used to determine susceptibility of H. pylori to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* People who have H. pylori sensitive to all antibiotics before therapy and and do not eradicate H. pylori after appropriate antibiotic therapy.

Exclusion Criteria:

* People who did not eradicate H. pylori because of primary resistance to antibiotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators invited people who were not able to eradicate H. pylori although at their first visit they had H. pylori sensitive to all antibiotics tested. At first visit all patients had stomach biopsy sample taken and H. pylori isolated and therapy prescribed. If they did not eradicate bacteria after 2 months they were again invited to control visit to define the problem and appropriate therapy prescribed. They were again invitation to control visit at the end of June 2010 to see the outcome of therapy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sequence type of H.pylori determined with MLST as a good evidence that people are infected with only one strain of H. pylori | Six months after first visit the strains from before/after therapy will be inspected with MLST to see if people have mixed strain infection.
  The investigators assume that people that are not able to eradicate infection with H. pylori although they have never been treated for such infection and they have taken appropriate therapy, have such problems because H. pylori is capable to escape from immune response. The investigators will define if patients have the same H. pylori sequence type through longer period and that such H. pylori is capable to develope resistance to clarithromycin very quickly.Such patients can eliminate H. pylori if we check the infection status more often and give them more suitable antibiotic therapy.
Sequence type of H.pylori determined with MLST as a good evidence that people are infected with only one strain of H. pylori | 9 months after first visit to see if people still have H. pylori due to insufficient immune response.
  The investigators assume that people that are not able to eradicate infection with H. pylori although they have never been treated for such infection and they have taken appropriate therapy, have such problems because H. pylori is capable to escape from immune response. The investigators will define if patients have the same H. pylori sequence type through longer period and that such H. pylori is capable to develope resistance to clarithromycin very quickly.Such patients can eliminate H. pylori if we check the infection status more often and give them more suitable antibiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alojz Ihan, MD. PhD, Study Director — Institute of mircobiology and immunology, Slovenia
Locations (1):
- Institute of microbiology and immunology, Ljubljana, Slovenia